CLINICAL TRIAL: NCT04267536
Title: UPwArds - Post Marketing Observational Study to Evaluate the Impact of CRP-Level on the Real World Effectiveness of UPadacitinib When Used in MonotherApy or in Combination With MTX in Patients With RheumatoiD ArthritiS
Brief Title: An Observational Study to Evaluate Impact of CRP-Level on Real World Effectiveness of Upadacitinib as Monotherapy or in Combination With MTX in Adult Participants With Rheumatoid Arthritis
Acronym: UPWARDS
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-078
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid Arthritis (RA); Upadacitinib; RINVOQ; Methotrexate (MTX); ABT-494; C-reactive protein (CRP)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants treated with upadacitinib monotherapy: Participants will receive upadacitinib for 12 months as prescribed by the physician
- Participants treated with upadacitinib in combination with MTX: Participants will receive upadacitinib in combination with MTX as prescribed by the physician for 12 months

SUMMARY:
Rheumatoid Arthritis (RA) is a chronic inflammatory disease causing pain, stiffness, swelling and loss of joint function. RA can reduce the ability to perform everyday tasks. This study assesses whether C-reactive protein (CRP)-level has an impact on achieving remission with upadacitinib when used alone or in combination with methotrexate (MTX). This study will also assess the reduction in pain, morning stiffness, fatigue, functionality, health status and impact of RA.

CRP is an indicator of inflammation and often used for disease activity monitoring during RA treatment. Upadacitinib is a Janus kinase (JAK) inhibitor indicated for the treatment of adults with moderately to severely active RA who have had an inadequate response or intolerance to methotrexate. This study has two groups - upadacitinib monotherapy and combination. Adult participants with moderate to severe RA will be enrolled. Around 500 participants will be enrolled in the study in multiple sites within Germany.

Participants will receive upadacitinib alone or in combination with MTX per their physicians' usual prescription. Individual data will be collected for 12 months.

No additional study-related tests will be conducted during the routine physician visits. Only data which are routinely collected during a regular visit will be utilized for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe active rheumatoid arthritis (RA) upon judgment of the treating physician.
* Swollen Joint Count (SJC) >= 3 of 28 joints of the Disease Activity Score (DAS)28.
* Measurement of C-Reactive Protein (CRP)-level at Baseline (BL) or <= 4 weeks prior to BL at a timepoint when the Prednisolone equivalent dose of Glucocorticoid treatment was <= 10 mg/day for at least 7 days.
* Upadacitinib treatment is indicated as per local Summary of Product characteristics (SmPC).
* Decision on the treatment with Upadacitinib was made prior to any decision to approach the patient to participate in this study.

Exclusion Criteria:

* Participants who cannot be treated with Upadacitinib according to the local Upadacitinib SmPC.
* Prior treatment with Upadacitinib.
* Treatment with Sarilumab or Tocilizumab within the last 8 weeks before the CRP level for inclusion was measured.
* Participants currently participating in interventional research.
* Participants who are unwilling or unable to complete the patient reported questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Participants with moderate to severe rheumatoid arthritis (RA)
Sampling Method: Non-Probability Sample
Enrollment: 534 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Remission | 6 Months
  Remission is defined as clinical disease activity index (CDAI) <=2.8

SECONDARY OUTCOMES:
Percentage of Participants Achieving Remission | Up to 12 Months
  Remission is defined as the disease activity score at 28 joints (DAS28)-C-Reactive protein (CRP)<2.6, DAS28- erythrocyte sedimentation rate (ESR)<2.6, simplified disease activity index (SDAI)<=3.3, CDAI<=2.8, Boolean.
Percentage of Participants Achieving Low Disease Activity (LDA) | Up to 12 Months
  LDA is defined as DAS28-CRP<3.2, DAS28-ESR<3.2, SDAI <=11, CDAI<=10
Mean Change From Baseline in CDAI | Up to 12 Months
  The CDAI is a validated measure of RA disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, global health assessed by the participant on a visual analogue scale (VAS) from 0 to 10 (cm), and global health assessed by an investigator on a visual analogue scale from 0 to 10 (cm) were included in the CDAI score. Scores on the CDAI range from 0 (lowest disease activity) to 76 (highest disease activity).
Mean Change From Baseline in SDAI | Up to 12 Months
  The SDAI is a validated measure of RA disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, global disease activity assessed by the participant on a visual analogue scale from 0 to 10 (cm) , global disease activity assessed by an investigator on a visual analogue scale from 0 to 10 (cm), and serum levels of C-reactive protein (mg/dL) were included in the SDAI score. Scores on the SDAI range from 0 (lowest disease activity) to 86 (highest disease activity).
Mean Change From Baseline in DAS28-CRP | Up to 12 Months
  The Disease Activity Score (DAS) 28 is a validated index of rheumatoid arthritis disease activity. Scores on the DAS28 range from 0 (lowest disease activity) to 10 (highest disease activity).
Mean Change From Baseline in DAS28-ESR | Up to 12 Months
  The Disease Activity Score (DAS) 28 is a validated index of rheumatoid arthritis disease activity. Scores on the DAS28 range from 0 (lowest disease activity) to 10 (highest disease activity).
Percentage of Participants Achieving Pain Reduction (Improvement by 30 %) | Up to 12 Months
  Improvement in pain reduction is assessed by numeric rating scale (NRS). The NRS of Pain sheet will be filled out in the office by participants at the designated visits.
Percentage of Participants Achieving Pain Reduction (Improvement by 50 %) | Up to 12 Months
  Improvement in pain reduction is assessed by numeric rating scale (NRS). The NRS of Pain sheet will be filled out in the office by participants at the designated visits.
Percentage of Participants Achieving Pain Reduction (Improvement by 70 %) | Up to 12 Months
  Improvement in pain reduction is assessed by numeric rating scale (NRS). The NRS of Pain sheet will be filled out in the office by participants at the designated visits.
Mean Change From Baseline in Pain | Up to 12 Months
  The NRS of Pain sheet will be filled out in the office by participants at the designated visits.
Percentage of Participants Achieving Fatigue Reduction (Improvement by 30 %) | Up to 12 Months
  Improvement in fatigue reduction is assessed by numeric rating scale (NRS). The NRS of fatigue sheet will be filled out in the office by participants at the designated visits.
Percentage of Participants Achieving Fatigue Reduction (Improvement by 50 %) | Up to 12 Months
  Improvement in fatigue reduction is assessed by numeric rating scale (NRS). The NRS of fatigue sheet will be filled out in the office by participants at the designated visits.
Percentage of Participants Achieving Fatigue Reduction (Improvement by 70 %) | Up to 12 Months
  Improvement in fatigue reduction is assessed by numeric rating scale (NRS). The NRS of fatigue sheet will be filled out in the office by participants at the designated visits.
Mean Change From Baseline in Fatigue | Up to 12 Months
  Change in Fatigue is assessed by numeric rating scale (NRS). The NRS of fatigue sheet will be filled out in the office by participants at the designated visits.
Change From Baseline in Rheumatoid Arthritis Impact of Disease (RAID) | Up to 12 Months
  RAID is a tool for assessment of disease activity purely based on a patient questionnaire.
Percentage of Participants Achieving RAID <= 3 | Up to 12 Months
  RAID is a tool for assessment of disease activity purely based on a patient questionnaire.
Percentage of Participants Achieving RAID > 3 and <=4 | Up to 12 Months
  RAID is a tool for assessment of disease activity purely based on a patient questionnaire.
Percentage of Participants Achieving RAID > 4 and <=6 | Up to 12 Months
  RAID is a tool for assessment of disease activity purely based on a patient questionnaire.
Percentage of Participants Achieving RAID > 6 | Up to 12 Months
  RAID is a tool for assessment of disease activity purely based on a patient questionnaire.
Change From Baseline in Morning Stiffness Severity | Up to 12 Months
  Morning stiffness severity was assessed by a numeric rating-scale (NRS). Participants rated the severity of morning stiffness during the past week from 0 to 10 with 0 representing "not severe" and 10 "very severe".
Change From Baseline in Morning Stiffness Duration | Up to 12 Months
  The duration of morning stiffness was reported by participants as the average daily length during the past week in minutes (from time of awaking to time of maximal improvement).
Change From Baseline in Functionality (FFbH) | Up to 12 Months
  A self-administered patient questionnaire used to assess patient function based on 18 questions. The numerically coded responses to the questions are added to provide a total patient score.
Change From Baseline in Patient Health Questionnaire (PHQ-9) | Up to 12 Months
  The PHQ-9 is a 9-item questionnaire for assessing the severity of depression. Each question is answered on a scale from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 27, where higher scores indicate more severe depression.
Percentage of Participants With Minimal Clinically Important Difference (MCID) in PHQ-9 | Up to 12 Months
  MCID is defined as the at least 5 points difference from baseline in PHQ-9. The PHQ-9 is a 9-item questionnaire for assessing the severity of depression.
Percentage of Participants With Low Disease Activity (LDA) or Remission Without Actual Concomitant MTX | Up to 12 Months
  LDA is defined as DAS28 < 3.2, CDAI<=10, SDAI <11. Remission is defined as DAS28<2.6, CDAI<=2.8; Boolean Remission.
Percentage of Participants With LDA or Remission With Actual Concomitant MTX | Up to 12 Months
  LDA is defined as DAS28 < 3.2, CDAI<=10, SDAI <11. Remission is defined as DAS28<2.6, CDAI<=2.8; Boolean Remission.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (52):
- Germany (52):
  - Praxis Dr. Rinaldi /ID# 218424, Ulm, Baden-Wurttemberg
  - Praxis Dres. Kellerer/Kellerer/Krüger /ID# 218428, Munich, Bavaria
  - Rheumahaus Studien GbR, Potsdam, DE /ID# 218430, Potsdam, Brandenburg
  - Rheumazentrum Ruhrgebiet /ID# 221388, Herne, North Rhine-Westphalia
  - Praxis Dr. Lüthke /ID# 218900, Dresden, Saxony
  - Kupka & Kupka, Altenburg, DE /ID# 218413, Altenburg
  - Marycz, Amberg, DE /ID# 220808, Amberg
  - Rheumapraxis am Webereck /ID# 218712, Augsburg
  - MVZ Weserbergland /ID# 220809, Bad Pyrmont
  - Internistische-rheumatologische Praxisgemeinschaft /ID# 218540, Bayreuth
  - Bozorg-Doagoo, Berlin, DE /ID# 218431, Berlin
  - Praxis Dr. Silke Zinke /ID# 218433, Berlin
  - Eisterhues, Braunschweig, DE /ID# 218532, Braunschweig
  - Medizinische Versorgungszentren Burghausen Altoetting /ID# 221385, Burghausen
  - Med Versorgungszentrum AGILOMED /ID# 218538, Chemnitz
  - Dres. Schuh /ID# 218541, Coburg
  - Rheumatologisches MVZ Dresden /ID# 218411, Dresden
  - Rheumapraxis Düren /ID# 224950, Düren
  - Strothmeyer & Scheulen /ID# 218426, Düsseldorf
  - Praxis Dilltal /ID# 218427, Ehringshausen
  - Praxisgemeinschaft Rheumatologie Nephrologie Erlangen /ID# 222579, Erlangen
  - Dres. Waehrisch/Flaxenberg /ID# 218711, Essen
  - Michael Mueller, Freiberg, DE /ID# 218414, Freiberg
  - Praxis Dr. Kuehne /ID# 221389, Haldensleben I
  - Praxis Dr. Liebhaber /ID# 218899, Halle
  - Aries, Hamburg, DE /ID# 220804, Hamburg
  - Stille, Hanover, DE /ID# 218429, Hanover
  - Medizinische Hochschule Hannover /ID# 222068, Hanover
  - Heilig, Heidelberg, DE /ID# 221391, Heidelberg
  - Praxis K. Pagel /ID# 218714, Hoppegarten
  - Hamann & Teich & Boche,Leipzig /ID# 218531, Leipzig
  - Schwarze/Haeder, Leipzig, DE /ID# 218412, Leipzig
  - Dres. Teipel/Toussaint/Saech /ID# 223969, Leverkusen
  - Aurich & Sieburg, Magdeburg /ID# 220811, Magdeburg
  - Harmuth, Marktredwitz, DE /ID# 218715, Marktredwitz
  - Prof-med-stud.de /ID# 218534, Munich
  - Praxis Dr. med Thilo Klopsch /ID# 218535, Neubrandenburg
  - Praxis Hein & Gess /ID# 218716, Nienburg
  - Praxis Hein & Gess /ID# 218896, Nienburg
  - Elisabeth-Klinik Bigge /ID# 218425, Olsberg
  - MVZ für Rheumatologie Dr. M. Welcker GmbH /ID# 218543, Planegg
  - Knappschaftsklinikum Saar /ID# 218901, Püttlingen
  - Rheumazentrum Ratingen /ID# 218897, Ratingen
  - Rheumatologische Gemeinschaftspraxis Schwerin /ID# 218432, Schwerin
  - Melzer, Seesen, DE /ID# 220803, Seesen
  - Rheumatologische Schwerpunktpraxis /ID# 218415, Stuttgart
  - Bruederkrankenhaus Trier /ID# 221393, Trier
  - Praxis Dr. Haas /ID# 218423, Tübingen
  - Rheumathologie Ulm /ID# 218539, Ulm
  - Krankenhaus St. Josef /ID# 221392, Wuppertal
  - Praxis Barmen /ID# 218895, Wuppertal
  - Fricke-Wagner, Zwickau, DE /ID# 218533, Zwickau

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P20-078&Latitude=&Longitude=&LocationName=#additional-resources-section